CLINICAL TRIAL: NCT06123975
Title: Study of the Role of Immunologic Factors in Adenomyosis Patients With Infertility
Brief Title: Adenomyosis Patients With Infertility and Immunological Factors
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LM2021242
Record Dates: First submitted 2023-08-16; First posted 2023-11-09 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2023-08

CONDITIONS: Adenomyosis
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood was collected on the day of embryo transfer. And if the pregnancy test was positive at 14 days after embryo transfer, peripheral blood was collected at 21 days after the transfer and every 2 weeks thereafter until 12 weeks of gestation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adenomyosis Cohort: Infertile patients with adenomyosis who met the inclusion and exclusion criteria, after signing the informed consent form, the researchers recorded the clinical information of the patients and initiated the IVF-ET procedure. Peripheral blood was collected on the day of embryo transfer. And if the pregnancy test was positive at 14 days after embryo transfer, peripheral blood was collected at 21 days after the transfer and every 2 weeks thereafter until 12 weeks of gestation.
  Interventions: Other: Venous blood collection

INTERVENTIONS:
Other: Venous blood collection — Peripheral blood was collected on the day of embryo transfer. And if the pregnancy test was positive at 14 days after embryo transfer, peripheral blood was collected at 21 days after the transfer and every 2 weeks thereafter until 12 weeks of gestation.

SUMMARY:
Infertile patients with adenomyosis who met the inclusion and exclusion criteria, after signing the informed consent form, the researchers recorded the clinical information of the patients and initiated the in vitro fertilization-embryo transfer (IVF-ET) procedure. Peripheral blood was collected on the day of embryo transfer. And if the pregnancy test was positive at 14 days after embryo transfer, peripheral blood was collected at 21 days after the transfer and every 2 weeks thereafter until 12 weeks of gestation. By analyzing the changes of immune cells and molecules in the peripheral blood of the patients, role of immune factors in infertility combined with adenomyosis was further explored.

DETAILED DESCRIPTION:
Adenomyosis is a common gynecological disease in women of reproductive age which is characterized by endometrial glands and stroma in the normal myometrium, accompanied by hypertrophy of the surrounding myometrial smooth muscle cells.The results of several studies showed that clinical pregnancy rate and live birth rate of in vitro fertilization-embryo transfer decreased in infertile patients with adenomyosis. This study intends to explore the immune-related mechanisms in infertile patients with uterine adenomyosis, with a view to finding effective clinical intervention targets for adenomyosis associated infertility, and providing new clues for the prevention and treatment of adenomyosis associated infertility. Peripheral blood was collected on the day of embryo transfer. And if the pregnancy test was positive at 14 days after embryo transfer, peripheral blood was collected at 21 days after the transfer and every 2 weeks thereafter until 12 weeks of gestation. The basic characteristics of the participants, such as age, body mass index, infertility type, infertility duration, gravida, parity times, basal follicle-stimulating hormone (FSH), anti-Müllerian hormone, uterine volume before IVF cycle, controlled ovulation hyperstimulation (COH) protocol, endometrial thickness, number of embryos transferred, transferred embryo type (cleavage embryo/blastocyst) were evaluated. Pregnancy outcomes of all patients were followed up. By analyzing the changes of immune cells and molecules in the peripheral blood of the patients, role of immune factors in infertility combined with adenomyosis was further explored.

ELIGIBILITY:
Inclusion Criteria:

* Patients were diagnosed as adenomyosis by transvaginal ultrasound scans (The criteria for sonographic diagnosis of adenomyosis are with 2 or more of the following: heterogeneous myometrial texture with the presence of globular asymmetric uterus, thickening of the anterior and posterior myometrial wall, irregular cystic areas within the myometrium);
* 18≤ age ≤ 40 years old at first outpatient visit in our Reproductive Center;
* with regular menstrual cycle.

Exclusion Criteria:

* Patients with intrauterine adhesion, uterine malformation, submucosal leiomyoma, or ≥ 5.0 cm in diameter leiomyoma;
* hydrosalpinx and systemic diseases;
* patients with other endocrine severe diseases, immune diseases, tumors and abnormal chromosomes in either partner.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile patients with adenomyosis who underwent IVF-ET at the Reproductive Center of the Peking University Third Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | Within 10 weeks after embryo transfer
  Clinical pregnancy denoted evidence of at least one intrauterine gestational sac observed by ultrasonography 30 days after embryo transfer. Clinical pregnancy rate = Number of patients who achieved clinical pregnancy / Number of transplant cycles.
Miscarriage rate | Within 24 weeks after embryo transfer
  Miscarriage was defined as the presence of an intrauterine gestational sac but no subsequent live birth after 24 weeks of gestation. Miscarriage rate = Number of patients with miscarriage / Number of patients who achieved clinical pregnancy.
Live birth rate | Within 1 year after embryo transfer
  Live birth was defined as delivery of a live baby after 24 weeks of gestation. Live birth rate = Number of patients with live birth / Number of transplant cycles.

SECONDARY OUTCOMES:
Immune cells and molecules in the peripheral blood | Within 12 weeks of gestation
  Immune cells and molecules in the peripheral blood on the day of embryo transfer, 21 days after the transfer and every 2 weeks thereafter until 12 weeks of gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Zhang, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No